CLINICAL TRIAL: NCT03294694
Title: A Phase 1 Study of the CDK4/6 Inhibitor Ribociclib (LEE011) in Combination With the PD-1 Inhibitor PDR001 in Patients With Metastatic Hormone Receptor-positive Breast Cancer and Metastatic Ovarian Cancer
Brief Title: Ribociclib + PDR001 in Breast Cancer and Ovarian Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Safety Implications
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Sara Tolaney, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-285
Record Dates: First submitted 2017-09-19; First posted 2017-09-27 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Hormone-Receptor-Positive (HR+) Breast Cancer; HER2-Negative Breast Cancer; Metastatic Epithelial Ovarian Cancer
Keywords: Metastatic Hormone-Receptor-Positive (HR+) Breast Cancer; HER2-Negative Breast Cancer; Metastatic Epithelial Ovarian Cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Ovarian Epithelial | interventions — ribociclib; spartalizumab; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ribociclib and PDR001 (Cohort A) (Experimental): * The treatment regimen is defined as ribociclib + PDR001.
  * Treatment will be administered on an outpatient basis.
  * The study will use a 3 + 3 dose escalation design to determine the MTD/RP2D.
  * Three to six evaluable patients will be enrolled in each cohort in the dose escalation phase.
    * Once the RP2D of the combination of ribociclib + PDR001 is determined, there will be an expansion cohort.
      * Cohort A expansion will assess the combination of ribociclib + PDR001 in 12 patients with metastatic ovarian cancer.
  Interventions: Drug: Ribociclib; Drug: PDR001
- Ribociclib, PDR001 and Fulvestrant (Cohort B) (Experimental): * The treatment regimen is defined as ribociclib + PDR001 + fulvestrant .
  * Treatment will be administered on an outpatient basis.
  * There will be a safety run-in using the MTD/RP2D of ribociclib + PDR001 from Cohort A with the addition of fulvestrant in an initial 6-12 patients.
    * Once the safety of the combination of ribociclib + PDR001 + fulvestrant is established, there will be an expansion cohort.
      * Cohort B expansion will assess the combination of ribociclib + PDR001 + fulvestrant in 24 patients with hormone receptor-positive metastatic breast cancer (HR+ MBC).
  Interventions: Drug: Ribociclib; Drug: PDR001; Drug: Fulvestrant

INTERVENTIONS:
Drug: Ribociclib — Each treatment cycle lasts 28 days. Ribociclib, 1 time per day by mouth for 21 days, followed by 1-week of rest (28-day cycle)
  Other Names: Kisqali; LEE011; LEE-011
Drug: PDR001 — Each treatment cycle lasts 28 days. (PDR001) will be administered once every 28 days (by intravenous infusion) over about 30 minutes (or up to 2 hours, if necessary) for the first infusion and over about 30 minutes for all following infusions.
Drug: Fulvestrant — Each treatment cycle lasts 28 days. Fulvestrant will be administered during Cycle 1 on days 1 and 15, and then on day 1 of each 28-day cycle thereafter.
  Other Names: Faslodex; ICI 182,780; ZD9238
  Arms: Ribociclib, PDR001 and Fulvestrant (Cohort B)

SUMMARY:
This clinical trial is studying the drug Ribociclib (LEE011) in combination with an immunotherapy drug called PDR001 (a therapy that uses the body's own immune system to control cancer) as a possible treatment for metastatic hormone-receptor-positive (HR+), HER2-negative breast cancer (in combination with fulvestrant) or metastatic epithelial ovarian cancer.

The names of the medications involved in this study are:

* Ribociclib (LEE011)
* PDR001
* Fulvestrant

DETAILED DESCRIPTION:
* This research study is a Phase I clinical trial, which tests the safety of an investigational combination of drugs (LEE011 with PDR001), and tries to define the appropriate dose of the above combination of investigational drugs to use for further studies. "Investigational" means that the intervention is being studied.
* The FDA (the U.S. Food and Drug Administration) has approved LEE011 as a treatment for hormone receptor positive metastatic breast cancer.
* The FDA has not approved PDR001 as treatment for any type of cancer.
* The FDA has approved fulvestrant as a treatment for hormone receptor positive metastatic breast cancer.
* When given separately these medications work in different ways to try and stop cancer cells from growing and spreading.

  * LEE011 is a drug designed to block certain proteins called cyclin-dependent kinases (CDKs) that are required for cells to divide. These proteins may also control the ability of certain cancers to grow.
  * PDR001 is an antibody. Antibodies are proteins usually produced by the body that help protect against foreign matter, such as bacteria and viruses. PDR001 blocks a protein called PD-1 which is present on cells called T-lymphocytes, which are involved in the immune response. PDR001 is being tested to see if it will allow the body's immune system to work against tumor cells. Other studies have shown that blocking PD-1 may result in reduced tumor cell growth in a variety of solid tumors.
  * Fulvestrant is an estrogen receptor antagonist that is indicated for the treatment of postmenopausal women with HR+ MBC.
* In this research study, the investigators are looking for a safe and tolerable dose of LEE011 that can be given in combination with PDR001 for participants with metastatic hormone-receptor-positive (HR+), HER2-negative breast cancer (in combination with fulvestrant) or metastatic epithelial ovarian cancer.

ELIGIBILITY FOR COHORT A DOSE ESCALATION (Ribociclib + PDR001):

* Hormone receptor (HR)-positive, HER2-negative metastatic breast cancer according to ASCO CAP Guidelines.

  * Participants may have received any number of previous endocrine/hormonal lines of therapy in the metastatic setting, as long as the last dose is ≥ 14 days prior to registration.
  * Participants may have received any number of prior lines of chemotherapy for advanced breast cancer as long as the last dose is ≥ 21 days prior to registration.
  * Prior therapy with biologics and investigational drugs is allowed as long as the last dose is ≥ 21 days prior to registration.
  * Prior CDK4/6 inhibition is allowed. Participants who have had prior ribociclib must have received treatment at full-dose without any dose-reductions. The last dose is required to be ≥ 21 days prior to registration
  * No prior PD1/PDL1/CTLA4 inhibitors
  * Participants may have received radiotherapy for palliative purposes but must have completed treatment ≥ 14 days prior to registration and not be experiencing > grade 1 treatment related toxicities.
  * Men are eligible, as long as on a GnRH agonist for at least 6 weeks prior to study entry. Men MUST remain on the GnRH agonist for the duration of protocol treatment.
  * Evaluable or measurable disease by RECIST 1.1.
* Metastatic epithelial ovarian cancer, fallopian tube or peritoneal cancer. All histologies (including serous, mucinous, endometrioid, clear cell, MMMTs and mix histologies) and tumor grades are eligible

  * Must have received a first-line platinum-based therapy and have disease that is platinum-resistant.

    --- Platinum-resistant disease is defined as disease relapse within 2 to 6 months of prior platinum-based chemotherapy.
  * There is no limit to the number of lines of prior chemotherapy, biology or hormonal therapy regimens.
  * No prior PD1/PDL1/CTLA4 inhibitors
  * Evaluable or measurable disease by RECIST 1.1.

ELIGIBILITY FOR COHORT A DOSE EXPANSION (Ribociclib + PDR001):

* Metastatic epithelial ovarian cancer, fallopian tube or peritoneal cancer. All histologies (including serous, mucinous, endometrioid, clear cell, MMMTs and mixed histologies) and tumor grades are eligible.

  * Must have received a first-line platinum-based chemotherapy regimen and have relapsed despite standard therapy.
  * Must have received a first-line platinum-based therapy and have disease that is platinum-resistant.

    --- Platinum-resistant disease is defined as disease relapse within 2 to 6 months of prior platinum-based chemotherapy.
  * There is no limit to the number of lines of prior chemotherapy, biology or hormonal therapy regimens.
  * Patients may have received any number of previous endocrine / hormonal lines of therapy in the metastatic setting, as long as the last dose is ≥ 14 days prior to first dose of study treatment.
* Prior therapy with biologics and investigational drugs is allowed, as long as the last dose is ≥ 21 days prior to first dose of study treatment.

  * No prior CDK4/6 inhibitors.
  * No prior PD1/PDL1/CTLA4 inhibitors.
  * Measurable disease by RECIST 1.1.
  * Participants with accessible tumor lesion(s) must be willing to undergo two research biopsies: one prior to treatment initiation and one after 7 weeks of protocol therapy. Participants who undergo an attempted on-treatment research biopsy and in whom inadequate tissue is obtained are still eligible to receive protocol therapy. They will not be required to undergo a repeat research biopsy attempt. If a biopsy-accessible participant has had a biopsy within 30 days of treatment initiation for clinical purposes, they may choose to submit an archived specimen from this procedure instead.

ELIGIBILITY FOR COHORT B SAFETY RUN-IN (Ribociclib + PDR001 + Fulvestrant):

* Hormone receptor (HR)-positive, HER2-negative metastatic breast cancer according to ASCO CAP Guidelines.
* Men are eligible, as long as on a GnRH agonist for at least 6 weeks prior to study entry. Men MUST remain on the GnRH agonist for the duration of protocol treatment.
* Women must be postmenopausal as defined as:

  -- Age >60 years or Age >45 with intact uterus and amenorrhea for >12 consecutive months or Follicle stimulating hormone (FSH) levels within postmenopausal range according to the ranges established by the testing facility or Premenopausal women who have been on a GnRH agonist for at least 6 weeks prior to study entry. Women in this group MUST remain on the GnRH agonist for the duration of protocol treatment or Status post bilateral oophorectomy, after adequate healing post-surgery
* Evaluable or measurable disease by RECIST 1.1.
* Prior CDK4/6 inhibition is allowed. Participants who have had prior ribociclib must have received treatment at full-dose without any dose-reductions. The last dose is required to be ≥ 21 days prior to registration
* Prior hormonal therapy:

  * Prior therapy with Fulvestrant is allowed
  * Participants may have received any number of previous endocrine/hormonal lines of therapy in the metastatic setting, as long as the last dose is ≥ 14 days prior to registration.
* Participants may have received chemotherapy for advanced breast cancer as long as the last dose is ≥ 21 days prior to registration.
* Prior therapy with biologics and investigational drugs is allowed as long as the last dose is ≥ 21 days prior to registration.
* Participants may have received radiotherapy for palliative purposes but must have completed treatment ≥ 14 days prior to registration and not be experiencing > grade 1 treatment related toxicities.

ELIGIBILITY FOR COHORT B DOSE EXPANSION (Ribociclib + PDR001 + Fulvestrant):

* Hormone receptor (HR)-positive, HER2-negative metastatic breast cancer according to ASCO CAP Guidelines.
* Men are eligible, as long as on a GnRH agonist for at least 6 weeks prior to study entry. Men MUST remain on the GnRH agonist for the duration of protocol treatment.
* Women must be postmenopausal as defined as:

  -- Age >60 years or Age >45 with intact uterus and amenorrhea for >12 consecutive months or Follicle stimulating hormone (FSH) levels within postmenopausal range according to the ranges established by the testing facility or Premenopausal women who have been on a GnRH agonist for at least 6 weeks prior to study entry. Women in this group MUST remain on the GnRH agonist for the duration of protocol treatment or Status post bilateral oophorectomy, after adequate healing post-surgery
* Prior hormonal therapy:

  * Participants may have received any number of previous endocrine/hormonal lines of therapy in the metastatic setting, as long as the last dose is ≥ 14 days prior to registration.
  * No prior fulvestrant
* Participants may have received up to one prior line of chemotherapy for advanced breast cancer as long as the last dose is ≥ 21 days prior to registration.
* Prior therapy with biologics and investigational drugs is allowed as long as the last dose is ≥ 21 days prior to registration.
* No prior CDK4/6 inhibitors
* No prior PD1/PDL1/CTLA4 inhibitors
* Participants may have received radiotherapy for palliative purposes but must have completed treatment ≥ 14 days prior to registration and not be experiencing > grade 1 treatment-related toxicities.
* Measurable disease by RECIST 1.1.
* Participants with accessible tumor lesion(s) must be willing to undergo two research biopsies: one prior to treatment initiation and one after 7 weeks of protocol therapy. Participants who undergo an attempted on-treatment research biopsy and in whom inadequate tissue is obtained are still eligible to receive protocol therapy. They will not be required to undergo a repeat research biopsy attempt. If a biopsy-accessible participant has had a biopsy within 30 days of treatment initiation for clinical purposes, they may choose to submit an archived specimen from this procedure instead.

ELIGIBILITY:
Inclusion Criteria

* Cohort A Dose Escalation (Ribociclib + PDR001) Eligibility can be found in Detailed Description Section
* Cohort B Safety Run-In (Ribociclib + PDR001 + Fulvestrant) Eligibility can be found in Detailed Description Section
* Cohort A Dose Expansion (Ribociclib + PDR001) Eligibility can be found in the Detailed Description Section
* Expansion Cohort B (Ribociclib + PDR001 + Fulvestrant Eligibility can be found in the Detailed Description Section
* ECOG Performance Status 0-1
* Participants must have normal organ and marrow function, as defined below:

  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * total hemoglobin ≥ 9 g/dL (may be post-transfusion)
  * total bilirubin ≤1.5 x institutional ULN (IULN)
  * AST(SGOT)/ALT(SGPT) ≤2.5 × IULN or ≤5 × IULN for participants with liver metastases
  * creatinine ≤1.5 x IULN or ≥ 60 ml/min/1.73m2 for subjects with creatinine levels above institutional normal
  * INR ≤ 1.5
  * estimated glomerular filtration rate (eGFR) ≥ 30 mL/min/1.73 by either Cockcroft-Gaultor CKD-EPI
  * baseline QTc ≤ 450 msec
* Age > 18 years
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, must be willing to use a highly effective method of contraception during dosing and for 150 days after the last dose of PDR001.

Note: Highly effective contraception methods include:

* Total abstinence (when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
* Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
* For female participants, male sterilization (at least 6 months prior to screening).
* Placement of an intrauterine device (IUD) or intrauterine system (IUS).

  * Sexually active males must be willing to use a condom during intercourse while taking the study drug and for 21 days after stopping the study drug and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.
  * Willingness to provide archival tumor samples. If sample is not available, a biopsy should be considered in patients with safely accessible disease. Participants who undergo an attempted research biopsy procedure for the purpose of this protocol, and in whom inadequate tissue is obtained, are not required to undergo repeat biopsy in order to continue on protocol.
  * Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants cannot have been treated on a prior interventional, investigational study within 2 weeks of the first dose of study treatment.
* Participants cannot receive treatment with any other investigational agents during protocol therapy.
* Use of hematopoietic colony-stimulating growth factors (e.g. G-CSF, GMCSF, M-CSF) ≤2 weeks prior start of study drug. An erythroid stimulating agent is allowed as long as it was initiated at least 2 weeks prior to the first dose of study treatment.
* History of severe hypersensitivity reactions to other mAbs
* Participants requiring chronic treatment with systemic steroid therapy, other than replacement-dose steroids in the setting of adrenal insufficiency within 7 days of treatment initiation. Topical, inhaled, nasal and ophthalmic steroids are allowed. Physiologic doses of steroids are acceptable.
* Participants receiving systemic treatment with any immunosuppressive medication (other than steroids as described above).
* Patient is currently receiving warfarin or other coumadin-derived anticoagulant for treatment, prophylaxis, or otherwise. Therapy with heparin, low molecular weight heparin (LMWH), coumadin or fondaparinux is allowed.
* Use of any live vaccines within 4 weeks of initiation of study treatment.
* Major surgery within 2 weeks of the first dose of study treatment (mediastinoscopy, insertion of a central venous access device, and insertion of a feeding tube are not considered major surgery).
* Participants with active autoimmune disease. Participants with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Presence of ≥ CTCAE grade 2 toxicity (CTCAE Grade 2 peripheral neuropathy and ototoxicity and any grade alopecia are allowed).
* Participants with uncontrolled intercurrent illness including, but not limited to:

  * Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormalities, including any of the following:

    * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis within 6 months prior to screening
    * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
    * Documented cardiomyopathy
    * Left Ventricular Ejection Fraction (LVEF) <50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO) within six months prior to beginning protocol therapy.
    * Clinically significant cardiac arrhythmias (e.g. ventricular tachycardia), complete left bundle branch block, high-grade AV block (e.g. bifascicular block, Mobitz type II and third-degree AV block)
    * Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome, or any of the following:
    * Risk factors for Torsades de Pointe (TdP) including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia.
    * Concomitant use of medication(s) with a known risk to prolong the QT interval and/or known to cause Torsades de Pointe that cannot be discontinued (within 5 half-lives or 7 days prior to starting study drug) or replaced by safe alternative medication
    * Systolic blood pressure (SBP) >160 mmHg or <90 mmHg at screening
    * Impairment of gastrointestinal function or who have gastrointestinal disease that may significantly alter the absorption of study drugs (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea or malabsorption syndrome).
    * Patient with liver disease and Child-Pugh score B or C.
  * Individuals with a history of a second malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and non-melanoma cancer of the skin. Patients with other cancers diagnosed within the past 5 years and felt to be at low risk of recurrence should be discussed with the study sponsor to determine eligibility.
  * Participants with known brain metastases may be enrolled in this study if radiation therapy and/or surgery have been completed with a minimum of 4 weeks of stable disease demonstrated on evaluation by MRI. Such participants must no longer require treatment with corticosteroids or enzyme inducing anti-epileptic medications for their CNS disease.
  * Participants with current pneumonitis.
  * Participants known to be HIV-positive or known to have active Hepatitis B or C.
  * Pregnant or lactating women. A negative pregnancy test in women of child-bearing potential must be documented within 7 days before the first dose of study medication.
  * Any condition that would prevent the patient's participation in the clinical study due to safety concerns, compliance with clinical study procedures or interpretation of study results.
  * Active infection requiring systemic antibiotic therapy.
  * Systemic anti-cancer therapy within 2 weeks of the first dose of study treatment. For cytotoxic agents that have major delayed toxicity, e.g. mitomycin C and nitrosoureas, 4 weeks is indicated as washout period. For patients receiving anticancer immunotherapies such as CTLA-4 antagonists, 3 weeks is indicated as the washout period
  * Participants who have received thoracic radiotherapy to lung fields ≤ 4 weeks prior to starting the study treatment or patients who have not recovered from radiotherapy-related toxicities. For all other anatomic sites (including radiotherapy to thoracic vertebrae and ribs) radiotherapy ≤ 2 weeks prior to starting the study treatment or has not recovered from radiotherapy-related toxicities. Palliative radiotherapy for bone lesions ≤ 2 weeks prior to starting study treatment is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2020-10-14 (Actual)

PRIMARY OUTCOMES:
Cohort A: MTD/RP2D of the Combination of Ribociclib + PDR001 | 4 weeks
  Toxicity will be graded according to NCI CTCAE, Version 4.0.
Cohort B: MTD/RP2D of the Combination of Ribociclib + PDR001 + Fulvestrant | 4 weeks
  Toxicity will be graded according to NCI CTCAE, Version 4.0.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | All participants will be evaluable for toxicity from the time of their first treatment with any study agent until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Toxicity will be graded according to NCI CTCAE, Version 4.0.
Objective Response Rate | 2 Years
  ORR is defined as the proportion of patients with complete response or partial response by RECIST 1.1 and immune-related RECIST (irRECIST)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Tolaney, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No